CLINICAL TRIAL: NCT00611260
Title: Does Meditation Improve Outcomes in Patients With Heart Failure Who Received Implantable Cardioverter Defibrillators and Cardiac Resynchronization Therapy Defibrillators?
Brief Title: Improvement in Clinical Outcomes in Heart Failure Patients With ICDs That Practice Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200715089
Record Dates: First submitted 2008-01-25; First posted 2008-02-08 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Congestive Heart Failure; Cardiac Resynchronization Therapy
Keywords: Meditation; Congestive Heart Failure; ICD; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure | interventions — Educational Status; Meditation; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meditation Cohort (Experimental): 25 patients will be given instruction in vipassana meditation. Vipassana meditation is thought to reduce the incidence of atrial and ventricular arrhythmias in patients with congestive heart failure, and improve their overall psychological profile.
  Interventions: Behavioral: Vipassana Meditation practice and instruction
- Standard Care (Active Comparator): 25 patients will receive current standard of care to manage their congestive heart failure, implanted cardiac devices, and psychological health.
  Interventions: Other: Standard Medical Care

INTERVENTIONS:
Behavioral: Vipassana Meditation practice and instruction — 2-3 instructed meditation sessions per week in addition to standard medical care.
  Other Names: Meditation + ICD
  Arms: Meditation Cohort
Other: Standard Medical Care — Standard medical care for patients with congestive heart failure plus implanted cardiac defibrillators.
  Other Names: Standard of Care
  Arms: Standard Care

SUMMARY:
This is a trial to examine the effects of meditation on the incidence of ventricular arrhythmias and the psychological profiles in patients with implanted cardiac defibrillators.

We wish to test the following hypotheses:

1. Vipassana meditation reduces the incidence of atrial and ventricular arrhythmias in patients with congestive heart failure.
2. Vipassana meditation improves the psychological profile in patients with CHF. In this study, subjects meeting the inclusion and exclusion criteria will be recruited into the study after obtaining informed consent. The subjects will then be randomized into either an experimental group ( Meditation) or into a control group (usual care).

DETAILED DESCRIPTION:
This is a single center, investigator-initiated, randomized, controlled trial to examine the effects of meditation on the incidence of ventricular arrhythmias and the psychological profiles in patients with implanted cardiac defibrillators and cardiac resynchronization devices. The former are used to protect patients against cardiac fibrillation and the latter for synchronizing the contractions of the two ventricles.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 85
* All patients with NYHA class II to III congestive heart failure symptoms from ischemic and non-ischemic etiology who received a defibrillator at least 3 months prior to enrollment.
* All patients with NYHA class III and IV symptoms, QRS complex of the ECG more than 120 ms, who received device for cardiac resynchronization at least 3 months prior to enrollment. These devices are placed when the two ventricles beat at slightly different times. These devices also have the capacity to record arrhythmias as the defibrillators.

Exclusion Criteria:

* Patients with life expectancy less than 6 months from non-cardiac causes
* Pregnant women
* Smokers
* History of major psychosis.
* Significant chronic liver, renal and pulmonary disease
* Active alcohol and drug abuse

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in ventricular arrhythmias and incidence of sudden cardiac death secondary to ventricular arrhythmias. | 3 month interval
Reduction of norepinephrine levels within the meditation assigned group resulting in improved quality of life. | 3 month intervals
Improved psychological profile of patients with CHF due to enhanced vitality and improved coping mechanisms resulting from participating in focused meditation. | 3 month intervals
Increase in heart rate variability for patients participating in vipassana meditation training. | 3 month intervals

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srivatsa, MD, Principal Investigator — University of California, Davis
Locations (1):
- UC Davis Medical Center, Sacramento, California, United States

REFERENCES:
- See also: Related Info — http://www.ucdmc.ucdavis.edu/clinicaltrials/trialDetail.aspx?protocol=200715089